CLINICAL TRIAL: NCT01827124
Title: Randomized Clinical Trial for Comparison Of Intravenous Carbeitocin Versus Oxytocin In Management Of Placental Delivery In Second Trimester Interruption
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wafaa Uthman Ahmed (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Sponsor-Investigator, Wafaa Uthman Ahmed, Ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: Ain Shams U
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-04

CONDITIONS: CARBETOCIN FOR PREVENTION OF PLACENTAL RETAINED
Keywords: CARBETOCIN AND OXYTOCIN AND SECOND TRIMESTER INTERRUPTION
MeSH Terms: interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carbetocin and placebo (Experimental): 100microgram carbetocin IV and 1cc normal saline(placebo)infusion
  Interventions: Drug: Carbetocin; Drug: oxytocin
- oxytocin and placebo (Experimental): 20Interntional unit oxytocin infusion and 1cc normal saline IV
  Interventions: Drug: Carbetocin; Drug: oxytocin

INTERVENTIONS:
Drug: Carbetocin
  Other Names: pabal
Drug: oxytocin
  Other Names: syntocinon

SUMMARY:
Intravenous Carbetocin is more efficient than intravenous infusion oxytocin in management of placental delivery in 2nd trimester interruption.

ELIGIBILITY:
Inclusion Criteria:

* Age:16-50 years
* Pregnancy duration: 14-24weeks
* Spontaneous abortion or medical induced abortion at 14-24weeks

Exclusion Criteria:

* Age less than 16years and more than 50 years
* Surgical termination
* Placenta previa
* Uterine fibroid

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Record duration of spontaneous placental expulsion after delivery of fetus in second trimester interruption | at the time of delivery

SECONDARY OUTCOMES:
Estimation of blood loss in each group by weighing all pads put under the patient after delivery of fetus tell expulsion of placenta( before and after using of pads). | at time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university maternity hospital department of obstetrics and gynacology, Cairo, Tertiary, Egypt